CLINICAL TRIAL: NCT01893177
Title: Open, Non-randomized Trial to Assess the Immunogenicity and Safety of the 2013/2014-season Virosomal Subunit Influenza Vaccine in Elderly and Young Subjects According to EMA Regulations
Brief Title: Re-licensing Study to Assess Inflexal V Formulated With WHO Recommended Influenza Strains (2013-14)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INF-V-A018
Record Dates: First submitted 2013-07-02; First posted 2013-07-08 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Influenza
Keywords: Influenza; Virus; Vaccination; Inflexal V
MeSH Terms: conditions — Influenza, Human; Virus Diseases | interventions — Inflexal V; Antigens, Surface; Virosomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elderly subjects aged over 60 years (Experimental)
  Interventions: Biological: Inflexal V
- Adults from 18 to 60 years old inclusive (Experimental)
  Interventions: Biological: Inflexal V

INTERVENTIONS:
Biological: Inflexal V — Intramuscular administration (M. deltoideus) of a single dose of 0.5 mL Inflexal V
  Other Names: Inflexal V influenza vaccine (surface antigen, inactivated, virosome) formulated for the WHO requirements of the 2013-2014 season, each 0.5 mL dose containing:; • 15 µg HA antigen of A/California/7/2009 (H1N1)-like virus; • 15 µg HA antigen of A/Texas/50/2012 (H3N2)-like virus; • 15 µg HA antigen of B/Massachusetts/2/2012-like virus

SUMMARY:
The study is to assess whether the influenza vaccine Inflexal V for season 2013/2014 fulfills the EMA requirements for re-registration of influenza vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male adults aged ≥18 on Day 1
* Written informed consent
* Female subjects of childbearing potential using and willing to continue using an acceptable method of contraception unless surgically sterilized/hysterectomized or post-menopausal for more than 2 years

Exclusion Criteria:

* Acute exacerbation of bronchopulmonary infection (cough, sputum, lung findings) or other acute disease
* Acute febrile illness (≥38.0 °C)
* Prior vaccination with an influenza vaccine in the past 330 days
* Known hypersensitivity to any vaccine component
* Previous history of a serious adverse reaction to influenza vaccine
* History of egg protein allergy or severe atopy
* Known blood coagulation disorder
* Chronic (longer than 14 days) administration of immunosuppressants or other immune-modifying drugs within 6 months before the first dose of the study vaccine, including oral corticosteroids in dosages of ≥0.5 mg/kg/d prednisolone or equivalent (inhaled or topical steroids are allowed)
* Known immunodeficiency (incl. leukemia, HIV seropositivity), cancer
* Investigational medicinal product received in the past 3 months (90 days)
* Treatment with immunoglobulins or blood transfusion(s) received in the past 3 months (90 days)
* Pregnancy or lactation
* Participation in another clinical trial
* Employee at the investigational site, or relative of the investigator
* Subjects who in the view of the investigator will not comply with study procedures and/or visit requirements as per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with seroconversion, seroprotection, and fold increase in geometric mean titer (GMT) | Day 22 +/- 2 days
  Immunogenicity variables are analyzed according to the EMA re-licensing criteria; at least one of the criteria has to be fulfilled for each vaccine strain:
  * Seroconversion rate at Day 22 has to be >40% of subjects aged ≥18 to ≤60 years and >30% of subjects aged >60 years, or
  * Seroprotection rate at Day 22 has to be >70% of subjects aged ≥18 to ≤60 years and >60% of subjects aged >60 years, or
  * GMT-fold increase at Day 22 compared to baseline: a >2.5-fold increase has to be reached in subjects aged ≥18 to ≤60 years and a >2.0-fold increase has to be reached in subjects aged >60 years

SECONDARY OUTCOMES:
Incidence of solicited local adverse events | Days 1 to 4 inclusive
Incidence of solicited systemic adverse events | Days 1 to 4 inclusive
Incidence of unsolicited adverse events | Days 1 to 22 inclusive

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, MD, Principal Investigator — Cross Research S.A.
Locations (1):
- CROSS Research S.A. - Phase I Unit, Arzo, Switzerland